CLINICAL TRIAL: NCT02476578
Title: Sending Advisory Electronic Mail to Primary Care Staff, Addressing Low Metabolic Measures: Assessing the Health Outcomes for Patients Above Age 75
Brief Title: Low Indexes of Metabolism - Information to Teams (LIMIT)
Acronym: LIMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Dr. Nir Tsabar, North District Principal Geriatrician, Clalit Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0023-15-COM; ר/2015/49 (Other Grant/Funding Number: The Israel National Institute for Health Policy Research); METABOL_EMAIL (Other: Clalit Health Organization North District Research Group); 0023-15-COM (Registry Identifier: Clalit Health Organization Community Division)
Record Dates: First submitted 2015-06-11; First posted 2015-06-19 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Weight Loss; Thinness; Malnutrition
Keywords: Hypocholesterolemia; Frail Elderly; Aged; Aged, 80 and over; Cholesterol; Clinical Laboratory Information Systems; Hemoglobin A, Glycosylated; diet therapy; Anticholesteremic Agents; Health Services for the Aged; Hypoglycemic Agents; Hypoglycemia
MeSH Terms: conditions — Weight Loss; Thinness; Malnutrition; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Email (Experimental): An email is sent, alerting the primary care providers about low values of BMI, HbA1c% or cholesterol and advising to consider appropriate dietary and medical revision.
  Interventions: Other: Email
- Control (No Intervention): No email is sent.

INTERVENTIONS:
Other: Email — Automated Email to the primary doctor and nurse, with the details of the patient, the condition found and the relevant measures to consider.
  Other Names: "Dry Counseling"
  Arms: Intervention Email

SUMMARY:
The purpose of this study is to determine whether alerting primary care providers by email about low values of BMI, HbA1c% or cholesterol will affect treatment and improve overall survival and other health indexes of people older than 75 years.

DETAILED DESCRIPTION:
Scientific background

Interventions aimed to ameliorate malnutrition are important for elderly health and include dietary counseling and discontinuing unnecessary medicines.

Emailing an alert regarding low BMI was found to improve dietary counseling numbers.

Correlation between death and HbA1c% is U-shaped, with increased mortality under a 6.5% level in patients taking two anti-diabetic medicines. Sending an email alert regarding an over-tight control of diabetes was followed by a reduction in mortality.

Death and cholesterol correlation is also U-shaped, with increased mortality and morbidity under 160 mg%. The investigator found no interventional study for this situation.

Objectives

To check whether alerting the primary care providers by email, about low values of BMI, HbA1c% or cholesterol will affect treatment and improve health indexes of people older than 75 years.

Working hypotheses

During a year, and relative to the control group, intervention emails may result in the following:

* A decrease in mortality.
* An increase in dietary counseling percentage and a decrease in prescribing anti-diabetic and cholesterol-lowering medicines.
* A decrease in medical expenses and in other morbidity indexes.

Type of research and methods of data collection

This randomized controlled trial will be conducted entirely through the existing computer system. The participants (patients) will be assigned to the two Arms/Groups "Intervention Email" and "Control". It has three separate interventions: a. Alerting about a significant drop in BMI. b. Alerting about a low HbA1c% level in patients taking anti-diabetics. c. Alerting about a low cholesterol level in patients taking cholesterol-lowering medicines. The alerts will be sent to the primary clinicians.

Method(s) of data analysis

Differences between intervention groups and control groups will be analyzed using Chi-square test (or Fishers' exact test) for categorical variables and using T-test (or Two-sample Wilcoxon test) for continuous variables.

Uniqueness and relevance

Health service policy regarding signs of malnutrition and excessive medicinal treatment needs a relevant scientific knowledge base. Nutritional counseling and revision of medicinal treatment may dramatically affect health. This research deals with questions that have no commercial interest, but are important to the public.

ELIGIBILITY:
Inclusion Criteria:

* All found by computerized search in the data base of Clalit Health Services North and South districts:
* 1. A drop in BMI of 2 Kg/m^2 or more during previous two years AND
* BMI less than 23 Kg/m^2 AND
* No dietitian counseling during previous year
* OR
* 2. Last HbA1c% level of 6.5% or less AND
* dispensing anti-diabetic medicines during previous 2 months
* OR
* 3. Last total cholesterol less than 160 mg/dL AND
* dispensing cholesterol-lowering medicines during previous 2 months

Exclusion Criteria:

* Patients whose their primary doctor and nurse email address is unobtainable
* For criterion 3: Patients diagnosed to have had a myocardial infarction, an ischemic heart disease, a transient ischemic attack or an ischemic stroke.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8584 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nir Tsabar, MD/PhD, Principal Investigator — ClalitHS North District Principal Geriatrist

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request to email nir.tsabar@clalit.org.il. Shared data will not include exact dates, exact lab results or any data that might expose the identity of patients. Also, commercial data such as drug brands or costs may not be shared.
Supporting Information: Study Protocol, SAP
Time Frame: After publishing the results in a peer reviewed journal.
Access Criteria: Any clinical researcher; Any ethically approved clinical research

REFERENCES:
- [Background] Flegal KM, Kit BK, Orpana H, Graubard BI. Association of all-cause mortality with overweight and obesity using standard body mass index categories: a systematic review and meta-analysis. JAMA. 2013 Jan 2;309(1):71-82. doi: 10.1001/jama.2012.113905. PMID 23280227
- [Background] Giovannelli J, Coevoet V, Vasseur C, Gheysens A, Basse B, Houyengah F. How can screening for malnutrition among hospitalized patients be improved? An automatic e-mail alert system when admitting previously malnourished patients. Clin Nutr. 2015 Oct;34(5):868-73. doi: 10.1016/j.clnu.2014.09.008. Epub 2014 Sep 18. PMID 25277380
- [Background] Iribarren C, Reed DM, Chen R, Yano K, Dwyer JH. Low serum cholesterol and mortality. Which is the cause and which is the effect? Circulation. 1995 Nov 1;92(9):2396-403. doi: 10.1161/01.cir.92.9.2396. PMID 7586337
- [Background] Currie CJ, Peters JR, Tynan A, Evans M, Heine RJ, Bracco OL, Zagar T, Poole CD. Survival as a function of HbA(1c) in people with type 2 diabetes: a retrospective cohort study. Lancet. 2010 Feb 6;375(9713):481-9. doi: 10.1016/S0140-6736(09)61969-3. Epub 2010 Jan 26. PMID 20110121
- [Result] Tsabar N, Press Y, Rotman J, Klein B, Grossman Y, Vainshtein-Tal M, Eilat-Tsanani S. A Randomized Trial of Alerting to Low Glycated Hemoglobin Level in Older Adults: Results of the Low Indexes of Metabolism Intervention Trial B (LIMIT-B). J Am Med Dir Assoc. 2020 Feb;21(2):277-280.e3. doi: 10.1016/j.jamda.2019.08.004. Epub 2019 Oct 3. PMID 31588026
- [Result] Tsabar N, Press Y, Rotman J, Klein B, Grossman Y, Vainshtein-Tal M, Eilat-Tsanani S. A Randomized Trial of Alerting to Hypocholesterolemia Results of the Low Indexes of Metabolism Intervention Trial-C (LIMIT-C). J Am Med Dir Assoc. 2020 Mar;21(3):410-414. doi: 10.1016/j.jamda.2019.08.018. Epub 2019 Oct 12. PMID 31610995
- [Result] Tsabar N, Press Y, Rotman J, Klein B, Grossman Y, Vainshtein-Tal M, Eilat-Tsanani S. Randomized trial results of alerting primary clinicians to severe weight loss among older adults in the Low Indexes of Metabolism Intervention Trial part A. Geriatr Gerontol Int. 2020 Apr;20(4):329-335. doi: 10.1111/ggi.13888. Epub 2020 Feb 16. PMID 32064727
- [Derived] Tsabar N, Press Y, Rotman J, Klein B, Grossman Y, Vainshtein-Tal M, Eilat-Tsanani S. The low indexes of metabolism intervention trial (LIMIT): design and baseline data of a randomized controlled clinical trial to evaluate how alerting primary care teams to low metabolic values, could affect the health of patients aged 75 or older. BMC Health Serv Res. 2018 Jan 5;18(1):4. doi: 10.1186/s12913-017-2812-0. PMID 29301522
- See also: Israel National Program for Quality Indicators in Community Healthcare — http://www.health.gov.il/Publicationsfiles/qindicatorsReport2008-2010.pdf
- Available data/document: Study Protocol — https://goo.gl/B6j1oF — LIMIT HEBREW PROTOCOL Version 3 (Final)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some of the participants may fit more than one criterion, as explained in the Eligibility section. Hence 7 subgroups are created:
  A) Fit only alert 1. B) Fit only alert 2. C) Fit only alert 3. D) Fit both alert 1. and alert 2. E) Fit both alert 1. and alert 3. F) Fit both alert 2. and alert 3. G) Fit all alerts: 1. , 2. and 3.
Period: Overall Study
Arm/Group | Intervention Email | Control
Started | 4310 | 4274
Died Before Email Was Sent (Died before 9.11.2015) | 35 | 43
Left Before End of Trial (Left district before 9.11.2016) | 6 | 13
Completed (Included in final analysis) | 4269 | 4218
Not Completed | 41 | 56
Not completed — Died before Email was sent (<9.11.2015) | 35 | 43
Not completed — Lost to Follow-up | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Email | Control | Total
Number analyzed (Participants) | 4269 | 4218 | 8487
Age, Continuous [Mean (Standard Deviation); unit: years] — Years old on 9.2015
  years | 80.6 (4.7) | 80.8 (4.9) | 80.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2484 | 2445 | 4929
  Male | 1785 | 1773 | 3558
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Israel | 4269 | 4218 | 8487
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (5.9) | 28.8 (5.9) | 28.8 (5.9)
HbA1c% Mean (Standard Deviation) [Mean (Standard Deviation); unit: %] — Population: Baseline HbA1c% in known for all participants in groups B,D,F,G. However, it is known only for some participants in groups A,C,E. (See: Eligibility section)
  %
    number analyzed (Participants) | 3185 | 3117 | 6302
    (all) | 6.51 (1.05) | 6.46 (1.00) | 6.49 (1.02)
Total Cholesterol Mean (Standard Deviation) [Mean (Standard Deviation); unit: mg/dL] — Population: Baseline Cholesterol is known for all participants in groups C,E,F,G. However, it is known only for some participants in groups A,B,D. See: Eligibility section.
  mg/dL
    number analyzed (Participants) | 4262 | 4209 | 8471
    (all) | 154.61 (33.88) | 154.23 (33.60) | 154.42 (33.74)

OUTCOME MEASURES:

1. Primary Outcome: Death From Any Cause
Description: Impact on overall-survival
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Email | Control
Number analyzed (Participants) | 4269 | 4218
Participants | 285 | 245

2. Secondary Outcome: Impact on Evaluation Rate
Description: Percentage of patients evaluated by a nurse and counseled by a dietitian
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Email | Control
Number analyzed (Participants) | 4269 | 4218
Participants | 3387 | 3337

3. Secondary Outcome: Impact on Medical Costs
Description: Medical expenses to the medical insurer, including hospitalizations, consultations, examinations, devices and medicines.
Time Frame: 1 year
Population: Data were not collected
Arm/Group | Intervention Email | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Impact on a Composite Measure of Medical Treatment
Description: A composite measure of doses of prescribed anti-diabetic and cholesterol-lowering medicines - According to relevant alert by email.
Time Frame: 1 year
Population: Data were not collected.
Arm/Group | Intervention Email | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 1 year
Description: Primary physicians and nurses who were recipients of the trial e-mail alert, were asked to report any adverse event to the principal investigator. No such report was received.
Arm/Group | Intervention Email | Control
All-Cause Mortality (participants affected / at risk) | 285/4269 | 245/4218
Serious Adverse Events (participants affected / at risk) | 0/4269 | 0/4218
Other Adverse Events (participants affected / at risk) | 0/4269 | 0/4218

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: APPROVED STUDY PROTOCOL, TRANSLATED FROM HEBREW (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT02476578/Prot_SAP_000.pdf